CLINICAL TRIAL: NCT01233297
Title: Antibiotic Treatment of Recurrent Episode of Asthma in Children - a Randomised, Case-controlled Study Within the COPSAC2010 Cohort (Asthma Begins in Childhood)
Brief Title: Antibiotic Treatment of Recurrent Episodes of Asthma in Children
Acronym: AB-studie
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Principal Investigator, Professor Klaus Bønnelykke, Professor, Copenhagen Studies on Asthma in Childhood
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-018592-16
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Childhood Asthma With Acute Exacerbation
Keywords: wheeze; infections
MeSH Terms: conditions — Respiratory Sounds; Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics (Active Comparator): Azithromycin (10 mg/kg once a day for 3 days)
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Placebo mixture (once a day for 3 days)
  Interventions: Other: Placebo mixture

INTERVENTIONS:
Drug: Azithromycin — 10 mg/kg peroral for 3 consecutive days
  Arms: Antibiotics
Other: Placebo mixture — Placebo mixture containing no active substance.
  Arms: Placebo

SUMMARY:
Copsac has discovered that asthmatic exacerbations are as closely linked to bacterial as to viral infection. The current study will examine whether treatment of asthmatic exacerbations with macrolide antibiotics - in the abscence of clear clinical bacterial infection which would in any case precipitate antibiotic treatment - has an effect on either the particular episode, or subsequently. Macrolide antibiotics are chosen for ease of administration ensuring high compliance, antibiotic appropriacy, and anti-inflammatory properties.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the COPSAC2010 cohort
* recurrent wheeze
* and others

Exclusion Criteria:

* Macrolide allergy
* Heart, liver or kidney disease.
* and others

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2010-11; Primary Completion 2027-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Symptom scoring | 1 to 3 years of age
Duration in days of each asthmatic episode from randomisation start | 1 to 3 years of age

SECONDARY OUTCOMES:
need for PO steroids during the episode | 1 to 3 years of age
beta-agonist use during the asthmatic episode | 1 to 3 years of age
time lapse until the next asthmatic episode | 1 to 3 years of age
MD assessment of the episode | 1 to 3 years of age
Family's assessment of the episode | 1 to 3 years of age
Asthma related health and economic assessment | 1 to 3 years of age
percentage of time away from kindergarten or, for the parents, away from work | 1 to 3 years of age
stratification of the above parameters according to bacterial colonisation of the airways | 1 to 3 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, MD, PhD, Principal Investigator — Copenhagen Studies on Asthma in Childhood
Locations (2):
- Denmark (2):
  - Copsac, DBAC, Gentofte Municipality, Copenhagen
  - Copsac, Næstved Hospital, Pediatric Department, Næstved

REFERENCES:
- [Derived] Mohammadzadeh P, Rosenberg JB, Vinding R, Mollegaard Jepsen JR, Lindberg U, Folsgaard N, Erlang Sorensen M, Sulaiman D, Bilenberg N, Mitta Raghava J, Fagerlund B, Vestergaard M, Pantelis C, Stokholm J, Chawes B, Larsson H, Glenthoj BY, Bonnelykke K, Ebdrup BH, Bisgaard H. Effects of prenatal nutrient supplementation and early life exposures on neurodevelopment at age 10: a randomised controlled trial - the COPSYCH study protocol. BMJ Open. 2022 Feb 1;12(2):e047706. doi: 10.1136/bmjopen-2020-047706. PMID 35105560
- [Derived] Thorsen J, Stokholm J, Rasmussen MA, Mortensen MS, Brejnrod AD, Hjelmso M, Shah S, Chawes B, Bonnelykke K, Sorensen SJ, Bisgaard H. The Airway Microbiota Modulates Effect of Azithromycin Treatment for Episodes of Recurrent Asthma-like Symptoms in Preschool Children: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2021 Jul 15;204(2):149-158. doi: 10.1164/rccm.202008-3226OC. PMID 33730519
- [Derived] Stokholm J, Chawes BL, Vissing NH, Bjarnadottir E, Pedersen TM, Vinding RK, Schoos AM, Wolsk HM, Thorsteinsdottir S, Hallas HW, Arianto L, Schjorring S, Krogfelt KA, Fischer TK, Pipper CB, Bonnelykke K, Bisgaard H. Azithromycin for episodes with asthma-like symptoms in young children aged 1-3 years: a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2016 Jan;4(1):19-26. doi: 10.1016/S2213-2600(15)00500-7. Epub 2015 Dec 17. PMID 26704020